CLINICAL TRIAL: NCT01791582
Title: Respiration Rate Parameter Studies in Healthy Volunteers Using a Bedside Respiratory Patient Monitoring System With the Multi-Functional Patient Monitoring PCBA-1
Brief Title: Pulse Oximetry- Evaluating Resp Rate- PCBA-1
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0304
Record Dates: First submitted 2012-11-29; First posted 2013-02-15 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess performance of resp rate parameter in a monitoring system PCBA-1

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 18 or older.
2. Subject is willing and able to provide written consent.

Exclusion Criteria:

1. Subject has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors.
2. Subjects with abnormalities that may prevent proper application of the device.
3. Subjects with significant Arrhythmia, as determined by subject self-report during screening and I/E criteria assessment at study start. (Three events of irregularities in radial pulse within thirty seconds).
4. Women who are pregnant or lactating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ME (mean error) of Respiration Rate values for each subject | 1-2 hours per subject

CONTACTS AND LOCATIONS:
Locations (1):
- Covidien, Boulder, Colorado, United States